CLINICAL TRIAL: NCT01251991
Title: Additive Cholesterol Lowering Effect by Concomitant Treatment With Psyllium Husks and Isolated Soy Protein in Addition to Heart-healthy Diet in Hypercholesterolemia
Brief Title: Cholesterol Lowering Treatment With Psyllium Husks and Isolated Soy Protein in Hypercholesterolemia
Acronym: ProFi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Anders Sorensen, Clinical dietitian, Aalborg University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2010-022822-34
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2011-06

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Soybean Proteins; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Combinatorial treatment (Experimental)
  Interventions: Drug: Psyllium husks; Dietary Supplement: Isolated soy protein
- Single treatment: Psyllium husks (Active Comparator)
  Interventions: Drug: Psyllium husks; Dietary Supplement: Isolated whey protein
- Single treatment: Isolated soy protein (Active Comparator)
  Interventions: Dietary Supplement: Isolated soy protein; Other: Microcrystalline cellulose
- Control (Placebo Comparator)
  Interventions: Dietary Supplement: Isolated whey protein; Other: Microcrystalline cellulose

INTERVENTIONS:
Drug: Psyllium husks — Oral suspension, oral use, two daily dosages consisting of 5 grams each
  Arms: Combinatorial treatment; Single treatment: Psyllium husks
Dietary Supplement: Isolated soy protein — Oral suspension, oral use, 30 grams once per day
  Arms: Combinatorial treatment; Single treatment: Isolated soy protein
Dietary Supplement: Isolated whey protein — Oral suspension, oral use, 30 grams once per day
  Arms: Control; Single treatment: Psyllium husks
Other: Microcrystalline cellulose — Oral suspension, oral use, two daily dosages consisting of 5 grams each
  Arms: Control; Single treatment: Isolated soy protein

SUMMARY:
Despite improved treatment, cardiovascular disease remains one of the most common diseases and causes of death in the Western world. Hypercholesterolemia is a well known risk factor for developing cardiovascular disease. Prevention and treatment are based in part on lowering LDL cholesterol. Dietary and lifestyle changes always play an important part of the treatment and preventive effort, and conversion to a heart-healthy diet reduces LDL cholesterol by a mean 10%. Further lowering of LDL cholesterol by means of food supplements have been demonstrated in numerous studies. Cholesterol lowering food supplements include isolated soy protein and water soluble dietary fibre such as psyllium husks. Postulated mechanisms of action responsible for the cholesterol lowering in these two food supplements are different, so there is a reason to expect an additive cholesterol lowering effect during concomitant treatment with both substances. The investigators want to investigate whether concomitant treatment with psyllium husks and isolated soy protein in addition to a heart-healthy diet results in a significantly greater reduction of LDL cholesterol in hypercholesterolemia, than single treatment with each of the substances.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18,5 - 35 kg/m2
* LDL cholesterol > 3,5 mmol/l

Exclusion Criteria:

* Triglycerides > 5,0 mmol/l
* Use of phytosterols, food supplements containing soy protein or water soluble fiber supplements
* Cardiovascular disease
* Diabetes mellitus
* Gastrointestinal disease
* Liver- og kidney disease
* Electrolyte imbalance
* Orlistat treatment
* Alcohol abuse
* Hypersensitivity to the interventional substances
* Pregnancy and nursing

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in LDL cholesterol at 6 weeks | 3rd and 4th visits at the investigational site
  3rd and 4th visits equal the ends of the 1st and 2nd intervention period at +6 weeks and +16 weeks from baseline respectively (4 week wash-out period in between the intervention periods). 2nd visit includes randomization and baseline measurement, while 1st visit @ -4 weeks compared to baseline includes screening and inclusion

SECONDARY OUTCOMES:
Change from baseline in total cholesterol at 6 weeks | 3rd and 4th visits at the investigational site
Change from baseline in HDL cholesterol at 6 weeks | 3rd and 4th visits at the investigational site
Change from baseline in triglycerides at 6 weeks | 3rd and 4th visits at the investigational site
Change from baseline in fasting plasma glucose at 6 weeks | 3rd and 4th visits at the investigational site
Change from baseline in body weight at 6 weeks | 3rd and 4th visits at the investigational site
Change from baseline in apolipoprotein B at 6 weeks | 3rd and 4th visits at the investigational site
Change from baseline in small, dense LDL cholesterol at 6 weeks | 3rd and 4th visits at the investigational site
Change from baseline in high sensitive CRP at 6 weeks | 3rd and 4th visits at the investigational site

CONTACTS AND LOCATIONS:
Overall Officials: Erik B. Schmidt, Professor, MD, Principal Investigator — Lipidklinikken, Aalborg Hospital
Locations (1):
- The Lipid Clinic, Aalborg Hospital, Aalborg, RN, Denmark